CLINICAL TRIAL: NCT02346734
Title: Physical Telerehabilitation in Veterans With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland (Other)
Collaborators: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Walter Royal, Director, Maryland Center for Multiple Sclerosis Treatment and Research, University of Maryland
Organization: University of Maryland, Baltimore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HP-00040344
Record Dates: First submitted 2014-05-07; First posted 2015-01-27 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Telerehablitation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSHAT (Active Comparator): The study participants will receive a clinical physical therapy evaluation and a physical therapy program to do at their own pace in the home and the intervention group will receive access to the MSHAT system via a website in which they will utilize each day. The study participants in the intervention group will login to the MSHAT system, go through a pre-exercise symptom diary to determine their eligibility to exercise, perform exercise while watching a video demonstration and report results real-time. The intervention group will also be able to send and receive messages via the MSHAT system. The time to complete the daily exercises will vary from patient to patient ranging for 10-30 minutes.
  Interventions: Device: Multiple Sclerosis Home Automated Telemanagement (MS HAT) system
- Control (No Intervention): The study participants randomized to group 2 will serve as the control. The study participants will receive a clinical physical therapy evaluation and a physical therapy program to do at their own pace in the home and will be given a paper diary to report their exercise completion. The control group will bring their paper diary showing their exercise completion results to their 3 month and 6 month follow-up visits.

INTERVENTIONS:
Device: Multiple Sclerosis Home Automated Telemanagement (MS HAT) system
  Arms: MSHAT

SUMMARY:
The primary objective of this study will be to assess the feasibility and patient acceptance of a Home Automated Telemanagement (HAT) system in multiple sclerosis patients.

Our hypothesis is that home telemanagement will be effective and useful in the rehabilitation of multiple sclerosis patients. Specifically, the investigators hypothesize that home telemanagement using a daily exercise diary, monitoring of compliance with a tailored exercise program and regular assessment of strength and motor functions will: 1. Be feasible and acceptable in patients with multiple sclerosis 2. Improve patient compliance with home exercise program 3. Increase patient mobility and motor functions 4. Be a feasible and effective mechanism for affecting multiple sclerosis patient self-efficacy 5. Improve quality of life

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65
* Clinical Diagnosis of MS based on McDonald criteria
* Functional disability defined by the PDDS in the range of 2 to 6
* Have a working telephone line in their home or a cell phone
* Willingness and ability to use MS HAT platform with individual modifications based on preferred user interface
* Patient demonstrates ability to successfully perform physical therapy exercises and procedures independently or with assistance of a caregiver.
* Ability to complete 25-foot walk test in at least 3 minutes

Exclusion Criteria:

* Age less than 18 years old
* No diagnosis of MS
* Other musculoskeletal diagnoses, unstable cardiovascular, respiratory, metabolic or other conditions that would interfere with this study
* One or more exacerbations in the preceding 3 months
* Received a course of steroids (IV or oral) within 60 days of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-07; Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
The Berg Balance Scale (BBS) | 6 month evaluation
  BBS consists of 14 activities common in daily life and is designed to measure balance in a clinical setting. The patient is asked to perform a task or to sustain a given position for a specific time. Points are deducted if the patient did not fulfill the time or activity requirements or touched an external support or received assistance from the examiner. Each item is rated from 0 to 4, 0 indicating the lowest level of function and 4 indicating the highest level of function. The total score sums up to 56. A score of 45 or above implies that an individual can safely move or walk independently.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | 6 month evaluation
  Expanded Disability Status Scale (EDSS) was developed for rating overall disability in MS. Patients are graded on the basis of presenting symptoms in eight different functional systems (FS), including pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, mental, and other functions. Scoring of the EDSS uses a 0 to 10, 20-step scale, with 0 equal to normal neurological function, 6.0 requires an assistive device for walking and 10.0 equal to death due to MS. The final score is based on grades obtained in the FS assessment.
9-Hole Peg Test | 6 month evaluation
  Measures finger dexterity
  * Administered by asking the patient to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible
  * Patients must then remove the pegs from the holes, one by one, and replace them back into the container
  * The board should be placed at the patient's midline, with the container holding the pegs oriented towards the hand being tested
  * Only the hand being evaluated should perform the test
  * Hand not being evaluated is permitted to hold the edge of the board in order to provide stability
  * Scores are based on the time taken to complete the test activity, recorded in seconds
  * Alternative scoring - the number of pegs placed in 50 or 100 seconds can be recorded. In this case, results are expressed as the number of pegs placed per second
  * Stopwatch should be started from the moment the participant touches the first peg until the moment the last peg hits the container
Paced Auditory Serial Addition Test | 6-month evaluation
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. It was developed by Gronwell in 1977 and later adapted by Rao and colleagues in 1989 for use in MS. The PASAT is presented using audio cassette tape or compact disk to ensure standardization in the rate of stimulus presentation. Single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it. Shorter inter-stimulus intervals, e.g., 2 seconds or less have also been used with the PASAT but tend to increase the difficulty of the task. Two alternate forms have been developed to minimize possible familiarity with the stimulus items when the PASAT is repeated over more than one occasion.
Patient Determined Disease Steps (PDDS) | 6-month evaluation
  The PDDS is a patient-reported outcome (PRO) of disability in multiple sclerosis. It has nine ordinal levels ranging between 0 (normal) to 8 (bedridden) and can be classified to mild, moderate and severe disability.
Range of motion | 6-month evaluation
  Range of motion refers to activity aimed at improving movement of a specific joint.
Lower extremities manual muscle test (LE-MMT) | 6-month evaluation
Functional Mobility | 6-month evaluation
Balance | 6-month evaluation
Gait | 6-month evaluation
Spasticity Scale (Modified Ashworth Scale) | 6-month evaluation
  Modified Ashworth Scale (MAS). MAS measures the resistance encountered during passive muscle stretching. Its scale ranges from 0 to 4: 0 = No increase in muscle tone; 1 = Slight increase in tone with a catch and release; 1+ = Slight increase in tone, manifested by a catch, followed by minimal resistance; 2 = Marked increase in tone; 3 = Considerable increase in tone; 4 = Rigid in flexion or extension.
Modified Fatigue Impact Scale (MFIS) | 6-month evaluation
  The Modified Fatigue Impact Scale (MFIS) is used to measure fatigue. The scale consists of 21 items, with 10 items related to mental fatigue, and 11 items relating to physical and social fatigue. The scoring ranges between 0 and 82, a high score reflecting greater impact. In the literature, a cut-off value of 38 has been used to discriminate fatigued from non-fatigued patients. It has shown good validity when compared with the Fatigue Severity Scale, but also appears to be more sensitive to the cognitive and psychosocial aspects of fatigue.
Multiple Sclerosis Walking Scale (MSWS-12) | 6-month evaluation
  MS Walking Scale (MSWS-12). MSWS-12 is a questionnaire with 12 items, measuring self-reported walking ability in MS. The questions are on limitations to patient's walking due to MS during the past 2 weeks. Each item ranges from 1 to 5 and the higher the sum, the more severe the degree of limitation.
MS Self-efficacy (MSSE) | 6-month evaluation
  MSSE is a 14-item questionnaire with a 6-point Likert scale, ranging from 1 (strongly disagree) to 6 (strongly agree). Self-efficacy is people's belief about their capabilities to overcome obstacles in life. Total score ranges from 14 to 84, a higher score indicating an elevated level of self-efficacy.
The Timed 25-Foot Walk (T25-FW) | 6-month Evaluation
  The patient is instructed to walk 25 feet as fast and as safely as possible. Then the patient repeats the task by walking back to the starting point. If necessary. assistive devices are allowed to be used. The amount of time (in seconds) that the patient took to walk 25 feet is measured.
The Six Minute Walk Test (6MWT) | 6-month evaluation
  The six minute walk test (6MWT) has been widely used as a measure of functional endurance in cadriopulmonary patients and is now being used as a practical and effective outcome measure to examine finctional exercise level in other chronic diseases including MS. Patients are asked to walk along a long, flat, straight, enclosed corridor with turnaround points marked with a cone.

OTHER OUTCOMES:
The Center for Epidemiologic Studies Depression Scale (CES-D) | 6-month evaluation
  The Center for Epidemiologic Studies Depression Scale (CES-D) will be used to measure depressive symptoms. CES-D is one of the most common screening tests for depression. This short self-administered test measures depressive feelings and behaviors during the past week. The scale includes 20 items and taps dimensions of depressed mood, feelings of guilt and worthlessness, appetite loss, sleep disturbance, and energy level. These items are assumed to represent the major components of depressive symptoms.
MOS Patient Adherence Measure | 6-month evaluation
  MOS Patient Adherence Measure is used to assess a patient's tendency to adhere to a doctor's recommendations during the past 4 weeks. Each item has a 6-point Likert Scale, ranging from 1 (none of the time) to 6 (all of the time). To score general adherence, the responses are averaged after reversing the items 1 and 3. By reversing the scores for items 1 and 3, overall positive aspects of patient adherence are measured.
Patient-Provider Communication (IPC) | 6-month evaluation
  Patients perceptions of their patient-provider communication quality will be measured using modified items from the Interpersonal Processes of Care (IPC) questionnaire. The IPC measures multiple facets of patient-provider communication such as general clarity, explanations of conditions and prognoses, and patients' preferences for various treatment options.
Syme's Social Networks Index (SNI) | 6-month evaluation
  Social networks will be measured by the widely used Berkman and Syme's Social Networks Index (SNI). The SNI assesses four types of social connections: marital (married or not); sociability (number and frequency of contacts with children, close relatives, and close friends); church group membership (yes versus no); and membership in other community organizations (yes versus no).

CONTACTS AND LOCATIONS:
Overall Officials: Walter Royal III, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States